CLINICAL TRIAL: NCT03373110
Title: Healthy Hearts Healthy Minds: A PPRN Demonstration Pragmatic Trial
Brief Title: Healthy Hearts Healthy Minds
Acronym: H3M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Andrew A. Nierenberg, MD, Director, Dauten Family Center for Bipolar Treatment Innovation, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017P001758
Record Dates: First submitted 2017-08-11; First posted 2017-12-14 (Actual); Results first posted 2021-04-29 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Cardiovascular Diseases; Depression
Keywords: Online Therapy; Fitbit; Depression; Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Online Mindfulness Based Cognitive Therapy +Fitbit (Experimental): A central aspect of MBCT is the concept of awareness. Participants practice a variety of meditation types (e.g. breath awareness) and learn to bring mindfulness to everyday situations. Awareness will be directed to elements in participants' lives that interfere with living a more productive, physically active life (e.g. thoughts and feelings that interfere with becoming more physically active; stressful situations and circumstances that prevent them from engaging in exercise). Two hundred participants will be randomized into this group.
  Interventions: Behavioral: Online Mindfulness Based Cognitive Therapy
- Online Cognitive Behavioral Therapy +Fitbit (Experimental): 1)identifying and setting realistic exercise-based goals and intermediate goals (to maximize success to increase motivation); (2) behavioral scheduling to optimize when to exercise, identify rewards for exercising, and problem solve obstacles to exercising; and (3) identify dysfunctional, maladaptive thoughts about exercise (which decrease motivation) and skills to identify more adaptive, positive thoughts (to overcome thoughts of being too tired or too stressed to exercise). Two hundred participants will be randomized into this group.
  Interventions: Behavioral: Online Cognitive Behavioral Therapy
- Fitbit Alone (Active Comparator): Participants assigned to the Fitbit-only control study group you will not be receiving therapy. However, they will receive a Fitbit, which they will be asked to wear over the course of 16 weeks as well as to complete the same schedule of assessments as the therapy arms. One hundred participants will be randomized into this group.
  Interventions: Behavioral: Fitbit Alone

INTERVENTIONS:
Behavioral: Online Mindfulness Based Cognitive Therapy — see arm description
  Arms: Online Mindfulness Based Cognitive Therapy +Fitbit
Behavioral: Online Cognitive Behavioral Therapy — see arm description
  Arms: Online Cognitive Behavioral Therapy +Fitbit
Behavioral: Fitbit Alone — see arm description
  Arms: Fitbit Alone

SUMMARY:
Healthy Hearts Healthy Minds: An Overview Individuals with depression are four times more likely to die from coronary heart disease than someone who does not have depression. At the same time, the risk of having a heart attack with depression is double that of individuals who do not have depression. Exercise, improves both depression and risk factors for heart disease; yet, most Americans do not exercise regularly, especially those with depression and/or heart disease.

This study is important to these individuals as most of them want to exercise, but have difficulty finding the motivation and energy to do so, which has a substantially negative impact on their physical and mental health. This study will compare two empirically supported treatments designed to help individuals with a mood disorder at risk or with heart disease to increase their physical activity as objectively measured by a Fitbit (which we will provide to participants at no cost).

This new study, focused on getting people moving, is funded by the Patient Centered Outcome Research Institute (PCORI) and involves 2 Patient Powered Research Networks (PPRNs) known as the MoodNetwork and the Health eHeart Alliance. With the help of patients across the country the Healthy Hearts Healthy Minds study team aims to be able to study the best method to get people to be more physically active - making them happier and healthier in the process.

DETAILED DESCRIPTION:
Healthy Hearts Healthy Minds: An Overview Individuals with depression are four times more likely to die from coronary heart disease than someone who does not have depression. At the same time, the risk of having a heart attack with depression is double that of individuals who do not have depression. Exercise, improves both depression and risk factors for heart disease; yet, most Americans do not exercise regularly, especially those with depression and/or heart disease.

This study is important to these individuals as most of them want to exercise, but have difficulty finding the motivation and energy to do so, which has a substantially negative impact on their physical and mental health. This study will compare two empirically supported treatments designed to help individuals with a mood disorder at risk or with heart disease to increase their physical activity as objectively measured by a Fitbit (which we will provide to participants at no cost).

This new study, focused on getting people moving, is funded by the Patient Centered Outcome Research Institute (PCORI) and involves 2 Patient Powered Research Networks (PPRNs) known as the MoodNetwork and the Health eHeart Alliance. With the help of patients across the country the Healthy Hearts Healthy Minds study team aims to be able to study the best method to get people to be more physically active - making them happier and healthier in the process.

What is the purpose of the study? Healthy Hearts Healthy Minds aims to compare two kinds of empirically supported treatment programs to see which is most effective at motivating people to be more physically active and increasing well-being: an online, standard, eight-week mindfulness training and an online, eight-session "cognitive-behavioral" training. The study may also tell us what groups of people do better with one or the other program.

How does the study work? 500 participants will be recruited from the MoodNetwork and the Health eHeart Alliance. They will be randomly assigned to either the mindfulness training, the cognitive-behavioral training, or a control group. Participants, regardless of group assignment, will receive a Fitbit Charge II at no cost.

All participants will fill out standard well-being and safety assessments every other week for eight weeks to see how they are doing. Participants will also do follow-up assessments after sixteen weeks has elapsed since starting the study. All sessions and assessments will be done online.

You may qualify if:

* You are physically active less than 150 minutes per week
* Have a body mass index (BMI) greater than 25kg/m2
* You possess an internet enabled device (e.g. smartphone, tablet/iPad, or desktop) with the Fitbit app and a registered personal account with Fitbit

What does participation involve?

* Wearing a FitBit Charge II throughout the duration of the 16 week study
* Filling out questionnaires via a secure, online system
* Potentially participating in additional weekly program sessions for 8 weeks, depending on which program you are assigned to.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give informed consent
* Fluent in English
* Between the ages of 18-65
* Lives in the United States
* Self-report of having experienced depression as assessed by the Mini International Neuropsychiatric Interview (MINI)
* Self report an elevated risk for or of having cardiovascular disease ( >150 minutes of physical activity a week)
* Registered a personal account with Fitbit prior to enrollment in the study

Exclusion Criteria:

* Unwilling/unable to comply with study procedures
* Pregnant
* Responds to item 9 (Suicidal ideation) on the PHQ-9 with a 3 or higher (i.e., "Thoughts that you would be better off dead or of hurting yourself in some way on more than half the days")
* Contraindications to exercise or diet interventions as assessed by the DASI
* Already uses a Fitbit device or other activity monitor
* Suffers from repeated episodes of "blacking out" or "fainting"
* Survived a cardiac arrest or sudden death
* Has recurrent chest discomfort with activity that goes away within 10 minutes of rest or with nitroglycerin
* Has heart failure
* Has been hospitalized recently (within past 6 weeks) for a cardiovascular problem

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dauten Family Center for Bipolar Treatment Innovation, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sylvia LG, Gold AK, Rakhilin M, Amado S, Modrow MF, Albury EA, George N, Peters AT, Selvaggi CA, Horick N, Rabideau DJ, Dohse H, Tovey RE, Turner JA, Schopfer DW, Pletcher MJ, Katz D, Deckersbach T, Nierenberg AA. Healthy hearts healthy minds: A randomized trial of online interventions to improve physical activity. J Psychosom Res. 2023 Jan;164:111110. doi: 10.1016/j.jpsychores.2022.111110. Epub 2022 Dec 1. PMID 36525851

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 491 participants were consented, 361 participants met eligibility criteria and were randomized to study intervention arms. 21 participants withdrew their consent and, thus, data from these 21 participants are not used or presented. Of the 340 randomized participants, 314 participants had usable Fitbit data. Therefore, 314 participants were included in all analyses (i.e., primary and secondary outcomes). We have added adverse event data on all randomized participants (i.e., 361 participants).
Period: Overall Study
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Started | 133 | 137 | 70
Provided Fitbit Data | 123 | 130 | 63
Completed | 55 | 58 | 26
Not Completed | 78 | 79 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone | Total
Number analyzed (Participants) | 133 | 137 | 70 | 340
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.5 (11.6) | 43.9 (11.2) | 43.4 (10.8) | 43.3 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 110 | 61 | 279
  Male | 25 | 27 | 9 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 12 | 5 | 26
  Not Hispanic or Latino | 122 | 124 | 64 | 310
  Unknown or Not Reported | 2 | 1 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 10 | 7 | 23
  White | 111 | 112 | 58 | 281
  More than one race | 11 | 10 | 3 | 24
  Unknown or Not Reported | 5 | 5 | 2 | 12
Bipolar Disorder [Count of Participants; unit: Participants] — Population: 3 participants were missing bipolar disorder diagnosis
  Participants
    number analyzed (Participants) | 132 | 136 | 69 | 337
    (all) | 18 | 21 | 12 | 51
Education [Count of Participants; unit: Participants]
  Some high school | 1 | 1 | 0 | 2
  High school graduate/GED | 8 | 9 | 8 | 25
  Some college/2-year degree | 43 | 50 | 21 | 114
  4-year college graduate | 31 | 37 | 14 | 82
  More than 4-year college | 49 | 39 | 27 | 115
  Missing/unknown | 1 | 1 | 0 | 2
Sexual Orientation [Count of Participants; unit: Participants]
  Straight | 103 | 118 | 54 | 275
  Lesbian | 4 | 1 | 5 | 10
  Gay | 5 | 2 | 2 | 9
  Bisexual | 5 | 11 | 6 | 22
  Asexual | 5 | 2 | 0 | 7
  Other | 7 | 1 | 2 | 10
  Missing/Unknown | 4 | 2 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change (Per Day) in Average Daily Steps From Baseline
Description: Participants randomized to the CBT+fitbit and MBCT+fitbit groups completed 8 weeks of online intervention sessions with biweekly questionnaires whereas participants in the fitbit only group completed 8 weeks of biweekly questionnaires alone. After the first 8 weeks of the study, participants received no new online intervention material (regardless of their initial group assignment), but were instructed to continue wearing their fitbit for the remaining 8 weeks of the study and the MBCT+fitbit and CBT+fitbit groups continued to have access to the intervention material presented in the first 8 weeks of the study. At week 16, participants completed a follow-up assessment. The Fitbit records start and stop times of the day (e.g., indicating when participants were in bed) and therefore, steps were only counted during these times. Participants without any step count data for a given day were treated as missing values for that day.
Time Frame: Baseline, 8 weeks, and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Average Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 123 | 130 | 63
Change (per day) in Average Daily Steps
  8 weeks | 2.8 [-1.7 to 7.0] | 2.9 [-1.3 to 7.0] | -8.2 [-14.5 to -1.9]
  16 weeks | -1.2 [-2.9 to 0.5] | -1.8 [-3.5 to -0.1] | -2.6 [-5.1 to -0.1]
Statistical Analysis 1: Comparison: Online Mindfulness Based Cognitive Therapy +Fitbit vs Online Cognitive Behavioral Therapy +Fitbit; We used linear mixed effects models fit via maximum likelihood to examine the effect of the interventions on daily steps. The models include a random intercept and fixed effects for intervention, time, and an intervention by time interaction. We used separate models to assess the intervention effects across the 8-week intervention period as well as the complete 16-week follow-up period; Test type: Other; p = 0.973, Mixed Models Analysis — A two-sided significance level of 0.05 was used for all analyses; The models include a random intercept and fixed effects for intervention, time, and an intervention by time interaction
Statistical Analysis 2: Comparison: Online Mindfulness Based Cognitive Therapy +Fitbit vs Fitbit Alone; We used linear mixed effects models to examine the effect of the interventions on average daily steps at 8 weeks into the study. These models account for the covariance of repeated measurements within subjects, and we used maximum likelihood estimation to adjust for missing daily step counts. The models include a random intercept and fixed effects for intervention, time, and an intervention by time interaction; Test type: Other; p = .005, Mixed Models Analysis — A two-sided significance level of 0.05 was used for all analyses; We used linear mixed effects models to examine the effect of the interventions on daily steps. These models account for the covariance of repeated measurements within subjects, and we used maximum likelihood estimation to account for missing daily step counts. The models include a random intercept and fixed effects for intervention, time, and an intervention by time interaction
Statistical Analysis 3: Comparison: Online Cognitive Behavioral Therapy +Fitbit vs Fitbit Alone; [analysis description as in outcome 1, analysis 2]; Test type: Other; p = .004, Mixed Models Analysis — A two-sided significance level of 0.05 was used for all analyses; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Online Mindfulness Based Cognitive Therapy +Fitbit vs Online Cognitive Behavioral Therapy +Fitbit; We used linear mixed effects models to examine the effect of the interventions on average daily steps at 16 weeks into the study. These models account for the covariance of repeated measurements within subjects, and we used maximum likelihood estimation to adjust for missing daily step counts. The models include a random intercept and fixed effects for intervention, time, and an intervention by time interaction; Test type: Other; p = 0.627, Mixed Models Analysis — A two-sided significance level of 0.05 was used for all analyses; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Online Mindfulness Based Cognitive Therapy +Fitbit vs Fitbit Alone; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.359, Mixed Models Analysis — A two-sided significance level of 0.05 was used for all analyses; [other analysis details as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Online Cognitive Behavioral Therapy +Fitbit vs Fitbit Alone; [analysis description as in outcome 1, analysis 4]; Test type: Other; p = 0.597, Mixed Models Analysis — A two-sided significance level of 0.05 was used for all analyses; [other analysis details as in outcome 1, analysis 2]

2. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by the Patient Health Questionnaire (PHQ-9)
Description: Change per day in average daily steps stratified by the Patient Health Questionnaire (PHQ-9). The PHQ-9 is a 9 item self-report measure assessing presence of depression. Individuals are asked to rank how often they have experienced each item over the past two weeks on a scale from 0 (not at all) - 3 (nearly every day). Possible total scores range from 0-27, with higher scores indicate higher levels of depression. The PHQ-9 is a continuous measure and thus, was left continuous in our model and was not categorized. Because the PHQ-9 is a continuous measure, we assumed a continuous linear change in the effect per unit change. For purposes of presenting the results, we selected scores of 5, 10, and 15 as values to report the model-based slopes.
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 123 | 130 | 63
Change (per day) in Avg Daily Steps
  8 weeks: PHQ-9 Score of 5 | 6.3 [.6 to 12.1] | 5.7 [-.2 to 11.6] | -9.1 [-17.4 to -.7]
  8 weeks: PHQ-9 Score of 10 | 3.0 [-1.3 to 7.2] | 3.2 [-.9 to 7.4] | -8.3 [-14.6 to -2.0]
  8 weeks: PHQ-9 Score of 15 | -.4 [-5.9 to 5.0] | .7 [-4.5 to 5.9] | -7.5 [-15.2 to .2]
  16 weeks: PHQ-9 Score of 5 | -1.1 [-3.4 to 1.2] | 0.9 [-1.5 to 3.2] | -2.2 [-5.5 to 1.1]
  16 weeks: PHQ-9 Score of 10 | -1.2 [-2.9 to 0.5] | -1.6 [-3.3 to 0.1] | -2.6 [-5.0 to -0.1]
  16 weeks: PHQ-9 Score of 15 | -1.3 [-3.5 to .9] | -4.1 [-6.4 to -1.9] | -2.9 [-6.0 to .1]

3. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by the Altman Self-Rating Mania Scale (ASRM)
Description: Change per day in average daily steps stratified by the Altman Self-Rating Mania Scale (ASRM), specifically using summed scores of 0,1, and 3. 5-item self rating scale, designed to asses the presence and/or severity of manic symptoms. Each item can be scored from 0-4. Possible total scores range from 0-25, and a score of 6 or higher indicates a high probability of a manic or hypomanic condition. The ASRM is a continuous measure and thus, was left continuous in our model and was not categorized. Because the ASRM is a continuous measure, we assumed a continuous linear change in the effect per unit change. For purposes of presenting the results, we selected scores of 0, 1, and 3 as values to report the model-based slopes.
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 123 | 130 | 63
Change (per day) in Avg Daily Steps
  8 week: ASRM score 0 | 2.6 [-2.8 to 8.0] | 3.1 [-2.3 to 8.6] | -11.6 [-19.1 to -4.1]
  8 week: ASRM score 1 | 2.7 [-1.8 to 7.2] | 3.0 [-1.5 to 7.6] | -9.9 [-16.6 to -3.3]
  8 week: ASRM score 3 | 2.9 [-1.9 to 7.7] | 2.8 [-1.6 to 7.2] | -6.6 [-13.2 to 0.0]
  16 week: ASRM score 0 | 0.3 [-1.9 to 2.5] | -.6 [-2.9 to 1.6] | -5.1 [-8.0 to -2.2]
  16 week: ASRM score 1 | -.5 [-2.4 to 1.3] | -1.2 [-3.1 to .7] | -3.9 [-6.5 to -1.3]
  16 week: ASRM score 3 | -2.2 [-4.1 to -0.2] | -2.3 [-4.1 to -.5] | -1.4 [-4.0 to 1.2]

4. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by the Well Being Index (WHO-5)
Description: Change per day in average daily steps stratified by the Well Being Index (WHO-5). 5 item self report measure (rated on a 6 point Likert scale) to assess quality of life. Possible total scores range from 0-100 with 0 representing worst possible quality of life and 100 representing best possible quality of life. The WHO-5 is a continuous measure and thus, was left continuous in our model and was not categorized. Because the WHO-5 is a continuous measure, we assumed a continuous linear change in the effect per unit change. For purposes of presenting the results, we selected scores of 15, 30, and 45 as values to report the model-based slopes.
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 133 | 137 | 70
Change (per day) in Avg Daily Steps
  8 weeks: WHO-5 score 15 | -1.4 [-7.2 to 4.4] | -1.3 [-6.9 to 4.3] | -10.2 [-17.5 to -2.9]
  8 weeks: WHO-5 score 30 | 2.2 [-2.1 to 6.6] | 2.5 [-1.7 to 6.6] | -8.0 [-14.3 to -1.7]
  8 weeks: WHO-5 score 45 | 5.8 [0.5 to 11.1] | 6.3 [1.1 to 11.4] | -5.9 [-13.6 to 1.9]
  16 weeks: WHO-5 score 15 | -2.0 [-4.4 to .4] | -3.5 [-5.8 to -1.2] | -3.9 [-6.8 to -1.0]
  16 weeks: WHO-5 score 30 | -1.4 [-3.1 to 0.4] | -2.0 [-3.8 to -0.3] | -2.5 [-5.0 to -.1]
  16 weeks: WHO-5 score 45 | -.7 [-2.8 to 1.5] | -.6 [-2.6 to 1.5] | -1.2 [-4.2 to 1.8]

5. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by the Perceived Stress Scale (PSS)
Description: Change per day in average daily steps stratified by the Perceived Stress Scale (PSS), specifically using scores of 15, 20, and 25. 10 item scale (rated 0-4) that aims to measure the degree to which situations in one's life are appraised as stressful. Possible total scores range from 0-40 with higher scores are associated with higher levels of perceived stress. The PSS is a continuous measure and thus, was left continuous in our model and was not categorized. Because the PSS is a continuous measure, we assumed a continuous linear change in the effect per unit change. For purposes of presenting the results, we selected scores of 15, 20, and 25 as values to report the model-based slopes.
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 123 | 130 | 63
Change (per day) in Avg Daily Steps
  8 weeks: PSS score 15 | 8.2 [2.2 to 14.3] | 6.3 [.2 to 12.4] | -4.8 [-13.2 to 3.6]
  8 weeks: PSS score 20 | 3.9 [-0.5 to 8.3] | 4.0 [-.4 to 8.4] | -7.2 [-13.7 to -.7]
  8 weeks: PSS score 25 | -.5 [-5.5 to 4.5] | 1.6 [-2.8 to 6.1] | -9.5 [-16.2 to -2.9]
  16 weeks: PSS score 15 | -.8 [-3.2 to 1.7] | -0.6 [-3.1 to 1.9] | -2.3 [-5.6 to 1.1]
  16 weeks: PSS score 20 | -1.1 [-2.9 to 0.5] | -1.5 [-3.2 to .3] | -2.5 [-5.1 to .1]
  16 weeks: PSS score 25 | -1.5 [-3.5 to 0.6] | -2.3 [-4.2 to -.4] | -2.7 [-5.4 to -.1]

6. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by Age
Description: Change per day in average daily steps stratified by age. Participants self-reported age on the demographics form. Age is a continuous measure and thus, was left continuous in our model and was not categorized. Because age is a continuous measure, we assumed a continuous linear change in the effect per unit change. For purposes of presenting the results, we selected ages of 35, 45, and 55 as values to report the model-based slopes.
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 123 | 130 | 63
Change (per day) in Avg Daily Steps
  8 weeks: age 35 | -2.8 [-8 to 2.5] | -2.2 [-7.6 to 3.2] | -2.5 [-10.3 to 5.4]
  8 weeks: age 45 | .6 [-3.9 to 5.0] | 3.3 [-.9 to 7.4] | -9.4 [-15.8 to -3.1]
  8 weeks: age 55 | 10.7 [4.6 to 16.8] | 8.7 [3.0 to 14.4] | -16.4 [-25.6 to -7.1]
  16 weeks: age 35 | -2.8 [-4.9 to -.8] | -2.6 [-4.9 to -0.4] | -2.0 [-5.1 to 1.2]
  16 weeks: age 45 | -1.8 [-3.5 to 0] | -1.8 [-3.5 to -.1] | -2.7 [-5.2 to -.2]
  16 weeks: age 55 | 1.5 [-1.1 to 4.1] | -.9 [-3.2 to 1.4] | -3.4 [-7 to .1]

7. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by Sex
Description: Change per day in average daily steps stratified by sex. Participants self-reported male or female on the demographics form.
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 123 | 130 | 63
Change (per day) in Avg Daily Steps
  8 weeks: Male | -1.9 [-11.8 to 8.0] | -10.7 [-20.6 to -.8] | -3.2 [-21.5 to 15.1]
  8 weeks: Female | 3.8 [-.9 to 8.6] | 5.8 [1.2 to 10.3] | -8.8 [-15.5 to -2.1]
  16 weeks: Male | 0.4 [-3.8 to 4.6] | -4.4 [-8.7 to -.1] | -12.0 [-20.4 to -3.7]
  16 weeks: Female | -1.5 [-3.4 to .4] | -1.3 [-3.1 to .6] | -1.7 [-4.3 to 0.9]

8. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by Anxiety
Description: Change per day in average daily steps stratified by anxiety. Comorbid anxiety was self-reported in the psychiatric history questionnaire.
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 133 | 137 | 70
Change (per day) in Avg Daily Steps
  8 weeks: Anxiety | -1.5 [-7.2 to 4.2] | 4.5 [-1.0 to 9.9] | -5.7 [-13.3 to 1.9]
  8 weeks: No anxiety | 9.6 [3.0 to 16.2] | .7 [-5.7 to 7.0] | -13.8 [-25.0 to -2.5]
  16 weeks: Anxiety | -1.8 [-4.1 to .4] | -3.6 [-5.9 to -1.4] | -.2 [-3.2 to 2.8]
  16 weeks: No anxiety | .7 [-2.0 to 3.4] | .7 [-1.9 to 3.2] | -7.7 [-12.0 to -3.4]

9. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by Smoking
Description: Change per day in average daily steps stratified by smoking status. Smoker or non-smoker was self-reported on the psychiatric history questionnaire.
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 133 | 137 | 70
Change (per day) in Avg Daily Steps
  8 weeks: Smoker | -18.2 [-39.6 to 3.2] | -17.3 [-34.4 to -.2] | -20.2 [-37.5 to -2.8]
  8 weeks: Non-smoker | 3.6 [-.8 to 8.0] | 4.1 [-.1 to 8.4] | -6.4 [-13.2 to .4]
  16 weeks: Smoker | -7.2 [-16.0 to 1.7] | -12.5 [-19.9 to -5.1] | -2.6 [-9.1 to 4.0]
  16 weeks: Non-smoker | -1.0 [-2.7 to 0.8] | -1.2 [-2.9 to .6] | -2.6 [-5.3 to .1]

10. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by Self-efficacy for Exercise (SEE)
Description: Change per day in average daily steps stratified by Self-efficacy for exercise (SEE), specifically using scores of 30, 45, and 55. Possible total scores range from 0-90. This 9-item measure, administered at study randomization, asks participants to indicate their self-confidence that they could exercise three times per week for twenty minutes under a variety of conditions. Sample items include being able to exercise if "You were bored by the program or activity" and "The weather was bothering you." Higher total scores on this measure reflect increased self-efficacy for exercise. The SEE is a continuous measure and thus, was left continuous in our model and was not categorized. Because the SEE is a continuous measure, we assumed a continuous linear change in the effect per unit change. For purposes of presenting the results, we selected scores of 30, 45, and 55 as values to report the model-based slopes.
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 133 | 137 | 70
Change (per day) in Avg Daily Steps
  8 week: SEE score 30 | 1.2 [-4.0 to 6.3] | 4.5 [-.1 to 9.9] | -6.0 [-13.3 to 1.2]
  8 week: SEE score 45 | 3.3 [-1.1 to 7.7] | 2.8 [-1.3 to 7.0] | -9.0 [-15.4 to -2.5]
  8 week: SEE score 55 | 4.7 [-.8 to 10.2] | 1.8 [-3.1 to 6.6] | -11.0 [-18.7 to -3.2]
  16 weeks: SEE score 30 | -1.0 [-3.1 to 1.1] | -.8 [-3.0 to 1.4] | -.3 [-3.1 to 2.6]
  16 weeks: SEE score 45 | -1.3 [-3.0 to .5] | -1.9 [-3.6 to -.2] | -3.4 [-5.9 to -.9]
  16 weeks: SEE score 55 | -1.4 [-3.6 to .8] | -2.5 [-4.5 to -.5] | -5.4 [-8.4 to -2.4]

11. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by the Duke Activity Status Index (DASI)
Description: Change (per day) in Average Daily Steps Stratified by the Duke Activity Status Index (DASI), specifically using summed scores of 40, 50, and 60. Possible total scores range from 0-58.2. This 12-item questionnaire, administered at the screening session, assesses an individual's current functional capabilities when engaging in various activities that involve physical exertion. Items include "Can you walk a block or two on level ground?" and "Can you climb a flight of stairs or walk up a hill?" Individual item responses are weighted based upon their metabolic cost, and subsequently summed to yield a total score. A higher score indicates better functional capability. The DASI is a continuous measure and thus, was left continuous in our model and was not categorized. Because the DASI is a continuous measure, we assumed a continuous linear change in the effect per unit change. For purposes of presenting the results, we selected scores of 40, 50, and 60 as values to report the model-based
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 133 | 137 | 70
Change (per day) in Avg Daily Steps
  8 week: DASI score 40 | 3.3 [-1.7 to 8.3] | 4.5 [-.7 to 9.6] | -7.6 [-14.7 to -.5]
  8 week: DASI score 50 | 2.6 [-1.8 to 7.0] | 2.4 [-1.8 to 6.6] | -8.4 [-15.0 to -1.8]
  8 week: DASI score 60 | 2.0 [-4.2 to 8.2] | .3 [-5.9 to 6.5] | -9.2 [-18.6 to .2]
  16 week: DASI score 40 | -2.0 [-4.0 to .1] | -1.9 [-4.0 to .2] | -3.5 [-6.2 to -.7]
  16 week: DASI score 50 | -1.0 [-2.7 to -.8] | -1.8 [-3.5 to 0.0] | -2.0 [-4.6 to .5]
  16 week: DASI score 60 | 0.0 [-2.4 to 2.5] | -1.6 [-4.2 to 1.0] | -.6 [-4.2 to 3.1]

12. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by the International Physical Activity Questionnaire (IPAQ) - Short Form
Description: Change (per day) in Average Daily Steps Stratified by the International Physical Activity Questionnaire (IPAQ) - Short Form, specifically at scores of 150, 350, and 850. This 7-item measure, administered at the screening and study randomization sessions, evaluates engagement in vigorous, moderate, and light (e.g., walking) activity in the prior 7 days. Higher scores on the IPAQ indicate higher activity levels. The IPAQ is a continuous measure and thus, was left continuous in our model and was not categorized. Because the IPAQ is a continuous measure, we assumed a continuous linear change in the effect per unit change. For purposes of presenting the results, we selected scores of 150, 350, and 850 as values to report the model-based slopes. We reported those values based on approximate 25th, 50th, 75th percentiles among baseline IPAQ scores among H3M participants.
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 133 | 137 | 70
Change (per day) in Avg Daily Steps
  8 week: IPAQ score 150 | 1.1 [-3.8 to 6.0] | 3.0 [-1.9 to 7.9] | -8.7 [-16.7 to -1.7]
  8 week: IPAQ score 350 | 2.0 [-2.8 to 6.8] | 2.9 [-1.9 to 7.7] | -9.8 [-17.4 to -2.2]
  8 week: IPAQ score 850 | 4.2 [-.4 to 8.9] | 2.7 [-1.9 to 7.2] | -12.5 [-19.8 to -5.1]
  16 week: IPAQ score 150 | -3.1 [-5.1 to -1.1] | -1.6 [-3.6 to .4] | -1.7 [-4.8 to 1.5]
  16 week: IPAQ score 350 | -2.8 [-4.7 to -.9] | -1.8 [-3.8 to .2] | -2.2 [-5.2 to .7]
  16 week: IPAQ score 850 | -2.2 [-4.0 to -.3] | -2.4 [-4.3 to -.5] | -3.6 [-6.5 to -.7]

13. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by Education
Description: Change (per day) in Average Daily Steps Stratified by education. Education was self-reported in the demographics questionnaire. Education is reported as: less than 4-year college, 4-year college, and more than 4-year college
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 133 | 137 | 70
Change (per day) in Avg Daily Steps
  8 weeks: less than 4 year college | -2.3 [-9.3 to 4.8] | -1.8 [-8.2 to 4.6] | -7.2 [-17.3 to 2.8]
  8 weeks: 4-year college | 2.1 [-6.9 to 11.1] | 5.5 [-2.2 to 13.1] | 9.3 [-5.9 to 24.5]
  8 weeks: more than 4-year college | 8.2 [1.3 to 15.0] | 7.4 [-.4 to 15.1] | -15.9 [-25.4 to -6.3]
  16 weeks: less than 4-year college | -.1 [-3.0 to 2.8] | -1.8 [-4.4 to .9] | -3.9 [-7.7 to 0.0]
  16 weeks: 4-year college | -4.9 [-8.5 to -1.3] | -2.4 [-5.7 to .9] | -4.2 [-10.0 to 1.5]
  16 weeks: more than 4-year college | .1 [-2.6 to 2.9] | -.9 [-3.9 to 2.1] | -.6 [-4.4 to 3.3]

14. Secondary Outcome: Change (Per Day) in Average Daily Steps Stratified by Employment
Description: Change (per day) in Average Daily Steps Stratified by the employment. Employment was self-reported in the demographics questionnaire. Employment is reported as employed, unemployed, and other.
Time Frame: Baseline, 8 and 16 weeks
Measure: Mean (95% Confidence Interval); unit: Change (per day) in Avg Daily Steps
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
Number analyzed (Participants) | 133 | 137 | 70
Change (per day) in Avg Daily Steps
  8 week: employed | 6.1 [.9 to 11.4] | 2.4 [-2.7 to 7.4] | -8.4 [-15.5 to -1.3]
  8 week: unemployed | -15.8 [-17.6 to -4.0] | 11.7 [0.2 to 23.3] | 2.8 [-21.8 to 27.5]
  8 week: other | 3.2 [-7.1 to 13.5] | -1.0 [-10.5 to 8.4] | -11.5 [-27.6 to 4.7]
  16 week: employed | .8 [-1.3 to 2.8] | -.6 [-2.7 to 1.5] | -2.1 [-5.0 to .8]
  16 week: unemployed | -14.9 [-19.7 to -10.0] | .5 [-4.2 to 5.2] | -2.6 [-11.7 to 6.5]
  16 week: other | 1.3 [-2.9 to 5.5] | -7.6 [-11.5 to -3.7] | -4.4 [-10.2 to 1.4]

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Data on adverse events were collected via a two-question survey designed to assess if participants have experienced any adverse events, related to the study, since starting to participate.
Arm/Group | Online Mindfulness Based Cognitive Therapy +Fitbit | Online Cognitive Behavioral Therapy +Fitbit | Fitbit Alone
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/145 | 0/72
Serious Adverse Events (participants affected / at risk) | 0/144 | 1/145 | 0/72
Other Adverse Events (participants affected / at risk) | 53/144 | 45/145 | 30/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Online Mindfulness Based Cognitive Therapy +Fitbit (N=144) | Online Cognitive Behavioral Therapy +Fitbit (N=145) | Fitbit Alone (N=72)
Angina (Cardiac disorders) | 0 (0) | 1 | 0 (0) — Hospitalized for Angina (coronary artery disease)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Online Mindfulness Based Cognitive Therapy +Fitbit (N=144) | Online Cognitive Behavioral Therapy +Fitbit (N=145) | Fitbit Alone (N=72)
Suicidal thoughts (Psychiatric disorders) | 43 | 39 | 23 — suicidal thoughts were not severe and were unrelated to the current study
Sleeping difficulty (Psychiatric disorders) | 0 | 0 | 1
Negative health event (Psychiatric disorders) | 7 | 5 | 5 — Event that caused disruption in ability to conduct normal life (not specified)
Hip injury (General disorders) | 1 | 0 | 0
Hospitalized for alcoholism (Psychiatric disorders) | 0 | 1 | 0
Cardiovascular procedure (Cardiac disorders) | 2 | 0 | 0 — Echocardiogram, cardiac stress test
Chronic kidney disease (General disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
(1) Our sample was disproportionately white (83%), female (82%), and highly educated (i.e., 92% had a college education or more); (2) study data (e.g., medical history, psychiatric diagnoses, mood symptoms, overall wellness) were self-report; and (3) we did not provide any personal contact with study staff for clarifying study procedures, supporting the intervention material, and/or troubleshooting technical issues with the Fitbit or online platform unless participants proactively emailed us.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/10/NCT03373110/Prot_SAP_000.pdf